CLINICAL TRIAL: NCT02885025
Title: Effects of Broccoli Sprout Extract on Allergic Rhinitis
Brief Title: Effects of Broccoli Sprout Extract on Allergy Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLNB-03-15F
Record Dates: First submitted 2016-08-23; First posted 2016-08-31 (Estimated); Results first posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-05

CONDITIONS: Rhinitis,Allergic
Keywords: hypersensitivity; antioxidants
MeSH Terms: conditions — Rhinitis, Allergic; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- BSE + Nasal Fluticasone (Active Comparator): subjects will be randomized into 1 of 4 arms:
  1. Broccoli Sprout Extract + Nasal Fluticasone
  2. Broccoli Sprout Extract + normal saline nasal spray
  3. Placebo Pill + Nasal Fluticasone
  4. Placebo Pill + normal saline nasal spray
  Interventions: Dietary Supplement: Broccoli Sprout Extract; Drug: fluticasone nasal
- Broccoli Sprout Extract + normal saline nasal spray (Active Comparator): subjects will be randomized into 1 of 4 arms:
  1. Broccoli Sprout Extract + Nasal Fluticasone
  2. Broccoli Sprout Extract + normal saline nasal spray
  3. Placebo Pill + Nasal Fluticasone
  4. Placebo Pill + normal saline nasal spray
  Interventions: Dietary Supplement: Broccoli Sprout Extract; Drug: normal saline nasal spray
- Placebo Pill + Nasal Fluticasone (Active Comparator): subjects will be randomized into 1 of 4 arms:
  1. Broccoli Sprout Extract + Nasal Fluticasone 2 Broccoli Sprout Extract + normal saline nasal spray 3. Placebo Pill + Nasal Fluticasone 4. Placebo Pill + normal saline nasal spray
  Interventions: Drug: fluticasone nasal; Dietary Supplement: broccoli sprout extract placebo
- Placebo Pill + normal saline nasal spray (Placebo Comparator): subjects will be randomized into 1 of 4 arms:
  1. Broccoli Sprout Extract + Nasal Fluticasone
  2. Broccoli Sprout Extract + normal saline nasal spray
  3. Placebo Pill + Nasal Fluticasone
  4. Placebo Pill + normal saline nasal spray
  Interventions: Dietary Supplement: broccoli sprout extract placebo; Drug: normal saline nasal spray

INTERVENTIONS:
Dietary Supplement: Broccoli Sprout Extract — Broccoli Sprout Extract contains the antioxidant Sulforaphane which is the active ingredient being studies.
  Arms: BSE + Nasal Fluticasone; Broccoli Sprout Extract + normal saline nasal spray
Drug: fluticasone nasal — fluticasone is a nasal steroid that is currently approved for treatment of allergic rhinitis.
  Arms: BSE + Nasal Fluticasone; Placebo Pill + Nasal Fluticasone
Dietary Supplement: broccoli sprout extract placebo — a tablet similar to the actual broccoli sprout extract though without BSE.
  Arms: Placebo Pill + Nasal Fluticasone; Placebo Pill + normal saline nasal spray
Drug: normal saline nasal spray — normal saline to replace nasal fluticasone in specific arms of the study
  Arms: Broccoli Sprout Extract + normal saline nasal spray; Placebo Pill + normal saline nasal spray

SUMMARY:
Allergic rhinitis is a common illness suffered among US Veterans. There are medications that help relieve allergy symptoms, including nasal steroid sprays and antihistamines. Some patients have increase symptoms with exposure to their trigger, such as a grasses when combined with pollution due to oxidative stress from pollution. In this study, patients with allergic rhinitis to grass will be given broccoli sprout extract that contains an antioxidant sulforaphane do see if there is beneficial effect in these patients.

DETAILED DESCRIPTION:
Allergic rhinitis is a common illness suffered among US Veterans. Despite the availability of medications, many patients fail to get adequate control of symptoms especially in high pollutant areas. Southern California air pollutants, like diesel exhaust particles may act as adjuvants to allergens leading to an exaggerated allergic response in certain individuals. These individuals may lack adequate Glutathione transferase activity; necessary to protect cells against pollutant induced oxidative stress. Sulforaphane has been shown to protect against oxidative stress. The investigators hypothesize consumption of foods containing high levels of sulforaphane are beneficial to US Veterans with GST deficiencies suffering from allergic rhinitis. In the investigators' preliminary data, the investigators discovered administration of broccoli sprout extract rich in sulforaphane leads to diminished nasal inflammatory reaction brought on by diesel exhaust particles though did not have sufficient patient numbers to prove an association with GST deficiency. The investigators propose a 3 week randomized clinical trial comparing broccoli sprout extract consumption with nasal corticosteroid administration after subjects with allergic rhinitis undergo a Timothy, Bermuda or Johnson grass nasal challenge. In Aims 1 and 2, the investigators will compare clinical (nasal symptom scores and peak nasal inspiratory flows) and laboratory (inflammatory cytokines, eosinophil cationic protein, tryptase) measurements between four groups: nasal corticosteroid, broccoli sprout extract, nasal corticosteroid plus broccoli sprout extract, and placebo. Aim 3 focuses on exploratory genetic analysis of the 3 glutathione S-transferase (GST) genes to determine if correlations exist between the inability to produce GST enzyme and the response to broccoli sprout extract. At the conclusion of this study, the investigators will gain further knowledge of which patients benefit from anti-oxidant nutritional supplementation in treating allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria

1. Females and males 18 years or older.
2. History consistent with seasonal allergic rhinitis consistent with grass allergy (symptoms during summer months, June through August, for at least two consecutive seasons).
3. Not currently taking any medications for allergic rhinitis.
4. Provide written informed consent.
5. Willing and able to comply with all aspects of the protocol.

Exclusion Criteria:

1. The subject has any uncontrolled or serious disease, or any medical or surgical or condition that in the opinion of the investigator(s) could affect the subject's safety and/or interfere with the study assessments.
2. History of anaphylaxis to environmental allergens or an unknown trigger.
3. History of broccoli allergy
4. Recent upper respiratory infection (less than 4 weeks prior to study) or other active Infection.
5. Active smoker
6. Currently receiving allergy immunotherapy.
7. History of rhinitis exacerbation within the past 2 weeks.
8. Use of non-selective Beta-Blocker.
9. Inability to give written informed consent.
10. History or evidence of non-stable cognitive capacity within less than 1 year (i.e. Alzheimer's disease, dementia, bipolar disorder) that in the opinion of the investigator(s) could affect the subject's safety and/or interfere with the study assessments.
11. Pregnancy
12. Perennial rhinitis
13. Uncontrolled asthma
14. Forced Expiratory Volume in 1 second <70% predicted at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA; Joseph Stephen Yusin, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the VA Greater Los Angeles Healthcare System Allergy Immunology Clinic
Groups:
- BSE + Nasal Fluticasone: subjects will be randomized into 1 of 4 arms:
  1. BSE + Nasal Fluticasone
  2. BSE + normal saline nasal spray
  3. Placebo Pill + Nasal Fluticasone
  4. Placebo Pill + normal saline nasal spray
  Broccoli Sprout Extract: Broccoli Sprout Extract contains the antioxidant Sulforaphane which is the active ingredient being studies.
  fluticasone nasal: fluticasone is a nasal steroid that is currently approved for treatment of allergic rhinitis.
- BSE + Normal Saline Nasal Spray: subjects will be randomized into 1 of 4 arms:
  1. BSE + Nasal Fluticasone
  2. BSE + normal saline nasal spray
  3. Placebo Pill + Nasal Fluticasone
  4. Placebo Pill + normal saline nasal spray
  Broccoli Sprout Extract: Broccoli Sprout Extract contains the antioxidant Sulforaphane which is the active ingredient being studies.
  normal saline nasal spray: normal saline to replace nasal fluticasone in specific arms of the study
- Placebo Pill + Nasal Fluticasone: subjects will be randomized into 1 of 4 arms:
  1. BSE + Nasal Fluticasone
  2. BSE + normal saline nasal spray
  3. Placebo Pill + Nasal Fluticasone
  4. Placebo Pill + normal saline nasal spray
  fluticasone nasal: fluticasone is a nasal steroid that is currently approved for treatment of allergic rhinitis.
  broccoli sprout extract placebo: a tablet similar to the actual broccoli sprout extract though without BSE.
- Placebo Pill + Normal Saline Nasal Spray: subjects will be randomized into 1 of 4 arms:
  1. BSE + Nasal Fluticasone
  2. BSE + normal saline nasal spray
  3. Placebo Pill + Nasal Fluticasone
  4. Placebo Pill + normal saline nasal spray
  broccoli sprout extract placebo: a tablet similar to the actual broccoli sprout extract though without BSE.
  normal saline nasal spray: normal saline to replace nasal fluticasone in specific arms of the study
Period: Overall Study
Arm/Group | BSE + Nasal Fluticasone | BSE + Normal Saline Nasal Spray | Placebo Pill + Nasal Fluticasone | Placebo Pill + Normal Saline Nasal Spray
Started | 16 | 14 | 9 | 8
Completed | 16 | 12 | 9 | 8
Not Completed | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 47 subjects had a positive reaction to the up dose grass allergen challenge that began with 75 subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | BSE + Nasal Fluticasone | BSE + Normal Saline Nasal Spray | Placebo Pill + Nasal Fluticasone | Placebo Pill + Normal Saline Nasal Spray | Total
Number analyzed (Participants) | 16 | 14 | 9 | 8 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 12 | 5 | 7 | 39
  >=65 years | 1 | 2 | 4 | 1 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 3 | 3 | 12
  Male | 12 | 12 | 6 | 5 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 1 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 1 | 3
  Black or African American | 4 | 5 | 4 | 4 | 17
  White | 7 | 8 | 3 | 3 | 21
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 14 | 9 | 8 | 47
PNIF [Mean (Standard Deviation); unit: L/min] — Peak Nasal Inspiratory Flow: Range is 0 - 400 L/min. Note that increase in value is consistent with decreased nasal resistance consistent with an improvement.
  L/min | 105 (21.2) | 120 (14.1) | 172.5 (31.8) | 170 (28.3) | 155 (49.5)

OUTCOME MEASURES:

1. Primary Outcome: Total Nasal Symptom Score (TNSS) Change From Baseline to 3 Weeks of Randomly Assigned Treatment
Description: The Immediate Total Nasal Symptom Score (TNSS): The TNSS has been used in prior interventional studies to evaluate different treatment modes for allergic rhinitis. The score will consist of subjects rating 4 symptoms (nasal congestion/postnasal drainage, nasal pruritus, rhinorrhea, or sneezing) on a scale of 0 to 3, where 0=no symptoms present, 1=mild symptoms that do not interfere with activity, 2=moderate symptoms that are slightly bothersome symptoms with slight interference with activity and/or nighttime sleep, or 3=severe symptoms with interference with activity and nighttime sleep. Thus minimal value would be 0 vs. maximal value would be a score of 12. A higher score correlates with higher rhinitis activity. Diminished scores following an intervention is consistent with an improvement in rhinitis symptoms.
Time Frame: measures at various points following challenge at baseline and 21 days
Population: intent to treat population (all participants assigned to 1 of the 4 groups above).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- BSE + Nasal Fluticasone: patients received combination of broccoli sprout extract tablet and nasal fluticasone for a total of 3 weeks
- BSE + Normal Saline Nasal Spray: Patients received broccoli sprout extract tablets and nasal saline spray for 3 weeks.
- Placebo Pill + Nasal Fluticasone: Patients received placebo tablet and nasal fluticasone for 3 weeks.
- Placebo Pill + Normal Saline Nasal Spray: Patients received placebo tablet and normal saline nasal spray for 3 weeks
Arm/Group | BSE + Nasal Fluticasone | BSE + Normal Saline Nasal Spray | Placebo Pill + Nasal Fluticasone | Placebo Pill + Normal Saline Nasal Spray
Number analyzed (Participants) | 16 | 12 | 9 | 8
score on a scale | -.5277 (0.1048) | -.5484 (.0014) | -.8359 (0.3903) | -.181 (.0846)

2. Primary Outcome: Peak Nasal Inspiratory Flow (PNIF) Change From Baseline to 3 Weeks of Randomly Assigned Treatment
Description: peak nasal inspiratory flow (PNIF) measures the peak flow during nasal inspiration with an approved device utilized in other studies. Measurements will be performed with TNSS (above).
Time Frame: 21 days (from randomization to completion)
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | BSE + Nasal Fluticasone | BSE + Normal Saline Nasal Spray | Placebo Pill + Nasal Fluticasone | Placebo Pill + Normal Saline Nasal Spray
Number analyzed (Participants) | 16 | 12 | 9 | 8
L/min | .3362 (.0026) | .1213 (.0607) | .0636 (.0485) | -.0538 (.0453)

3. Secondary Outcome: Interleukin 5 (IL5)
Description: Interleukin 5 (IL5) is considered a T2 cytokine that increases with exacerbations of atopic disease, including allergic rhinitis. Cytokine measurements are in pg/ml. Values are recorded with log transformation. Note that measurements are on a continuous score. Lower values are consistent with less T2 inflammation which is consistent with diminished or lower atopic/allergic response.
Time Frame: 21 days (from randomization to completion)
Measure: Mean (Standard Deviation); unit: log(pg/ml)
Arm/Group | BSE + Nasal Fluticasone | BSE + Normal Saline Nasal Spray | Placebo Pill + Nasal Fluticasone | Placebo Pill + Normal Saline Nasal Spray
Number analyzed (Participants) | 16 | 12 | 9 | 8
log(pg/ml) | -.5285 (.2236) | -.3213 (.2005) | -.1082 (.0083) | -.3755 (0.1866)

4. Secondary Outcome: Interleukin 4 (IL4)
Description: Interleukin 4 (IL4) is considered a T2 cytokine that increases with exacerbations of atopic disease, including allergic rhinitis. Cytokine measurements are in pg/ml. Values are recorded with log transformation. Note that measurements are on a continuous score. Lower values are consistent with less T2 inflammation which is consistent with diminished or lower atopic/allergic response.
Time Frame: 21 days (from randomization to completion)
Population: Patient diagnosed with grass induced allergic rhinitis were randomized into 1 of 4 groups.
Measure: Mean (Standard Deviation); unit: log(pg/ml)
Arm/Group | BSE + Nasal Fluticasone | BSE + Normal Saline Nasal Spray | Placebo Pill + Nasal Fluticasone | Placebo Pill + Normal Saline Nasal Spray
Number analyzed (Participants) | 16 | 12 | 9 | 8
log(pg/ml) | -.5655 (0.4738) | -.1076 (.0228) | -.3682 (.0294) | -.3695 (.233)

5. Secondary Outcome: Interleukin 6 (IL6)
Description: Interleukin 6 is a cytokine present during inflammatory process. This is recorded in pg/ml. Below is the log transformation of the pg/ml unit. Note that measurements are on a continuous score. Lower values are consistent with less inflammation which could occur with an inflammatory response.
Time Frame: 21 days (from randomization to completion)
Measure: Mean (Standard Deviation); unit: log(pg/ml)
Arm/Group | BSE + Nasal Fluticasone | BSE + Normal Saline Nasal Spray | Placebo Pill + Nasal Fluticasone | Placebo Pill + Normal Saline Nasal Spray
Number analyzed (Participants) | 16 | 12 | 9 | 8
log(pg/ml) | -1.0868 (.2903) | -.0519 (.2437) | -.2719 (1.6894) | .3567 (.2826)

6. Secondary Outcome: Interleukin 8 (IL8)
Description: Interleukin 8 s a cytokine that will increase with inflammation. Below is the log transformation of the pg/ml unit. Note that measurements are on a continuous score. Lower values are consistent with less inflammation which could occur with an inflammatory response.
Time Frame: 21 days (from randomization to completion)
Measure: Mean (Standard Deviation); unit: pg/ml log transformation
Arm/Group | BSE + Nasal Fluticasone | BSE + Normal Saline Nasal Spray | Placebo Pill + Nasal Fluticasone | Placebo Pill + Normal Saline Nasal Spray
Number analyzed (Participants) | 16 | 12 | 9 | 8
pg/ml log transformation | -.7626 (.0168) | -.047 (.0033) | -.1013 (.2629) | .0472 (.1748)

7. Secondary Outcome: Interleukin 13 (IL13)
Description: Interleukin 13 (IL13) is considered a T2 cytokine that increases with exacerbations of atopic disease, including allergic rhinitis. Cytokine measurements are in pg/ml. Values are recorded with log transformation. Note that measurements are on a continuous score. Lower values are consistent with less T2 inflammation which is consistent with diminished or lower atopic/allergic response.
Time Frame: 21 days (from randomization to completion)
Population: Patient diagnosed with grass induced allergic rhinitis were randomized into 1 of 4 groups.
Measure: Mean (Standard Deviation); unit: log(pg/ml)
Arm/Group | BSE + Nasal Fluticasone | BSE + Normal Saline Nasal Spray | Placebo Pill + Nasal Fluticasone | Placebo Pill + Normal Saline Nasal Spray
Number analyzed (Participants) | 16 | 12 | 9 | 8
log(pg/ml) | -1.0822 (.2568) | -.2985 (.0466) | .1577 (.1042) | -.0459 (.3745)

8. Secondary Outcome: Interleukin 1 Beta (IL1b)
Description: IL1b is a cytokine that will increase with inflammation. Below is the log transformation of the pg/ml unit. Note that measurements are on a continuous score. Lower values are consistent with less inflammation which could occur with an inflammatory response.
Time Frame: 21 days (from randomization to completion)
Population: Patient diagnosed with grass induced allergic rhinitis were randomized into 1 of 4 groups
Measure: Mean (Standard Deviation); unit: pg/ml with log transformation
Arm/Group | BSE + Nasal Fluticasone | BSE + Normal Saline Nasal Spray | Placebo Pill + Nasal Fluticasone | Placebo Pill + Normal Saline Nasal Spray
Number analyzed (Participants) | 16 | 12 | 9 | 8
pg/ml with log transformation | -.4058 (.2563) | .0183 (.037) | -.2382 (.3013) | .0713 (.1139)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study. 1 year 6 months total.
Description: Intermittent sneezing, expected adverse event. Flatulence, expected adverse event General: "cold like symptoms", unrelated, expected given time of year
  Nasal irritation after nasal saline spray, unrelated, unexpected :
  GI: hemorrhoids: unexpected, unrelated Chest pain: secondary to rib injury: unrelated, unexpected GI: bloating: expected
Groups:
- BSE + Nasal Fluticasone: subjects will be randomized into 1 of 4 arms:
  1. BSE + Nasal Fluticasone
  2. BSE + normal saline nasal spray
  3. Placebo Pill + Nasal Fluticasone
  4. Placebo Pill + normal saline nasal spray
  Broccoli Sprout Extract: Broccoli Sprout Extract contains the antioxidant Sulforaphane which is the active ingredient being studies.
  no adverse events reported fluticasone nasal: fluticasone is a nasal steroid that is currently approved for treatment of allergic rhinitis.
Arm/Group | BSE + Nasal Fluticasone | BSE + Normal Saline Nasal Spray | Placebo Pill + Nasal Fluticasone | Placebo Pill + Normal Saline Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 3/16 | 4/14 | 0/9 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BSE + Nasal Fluticasone (N=16) | BSE + Normal Saline Nasal Spray (N=14) | Placebo Pill + Nasal Fluticasone (N=9) | Placebo Pill + Normal Saline Nasal Spray (N=8)
gi complaints (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) — Flatulence
nasal symptom (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — sneezing
costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 | 0 | 1 (1) — patient went to ER during study for check pain that was reproducible and diagnosed with costochondritis
gi complaint (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 — hemorrhoids
viral urti (General disorders) | 1 (1) | 0 | 0 | 0 — viral upper respiratory track infection (nasal congestion, sneezing and rhinorrhea)
nasal irritation (General disorders) | 0 | 1 (1) | 0 | 0 — nasal irritation
abdominal bloating (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 — abdominal bloating
diarrhea (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 — diarrhea
nausea (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 — nausea

LIMITATIONS AND CAVEATS:
1. Difficult recruiting enough patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT02885025/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT02885025/ICF_001.pdf